CLINICAL TRIAL: NCT05457270
Title: A Randomized, Single-dose, Open-label, Single-center, Crossover Study to Assess the Relative Bioavailability and Safety of Different Formulations of AZD4831 in Fasted State in Healthy Volunteers.
Brief Title: A Study to Assess the Relative Bioavailability and Safety of Different Formulations of AZD4831 in Fasted State in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6580C00016
Record Dates: First submitted 2022-07-11; First posted 2022-07-13 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Healthy Volunteers
Keywords: Relative Bioavailability; AZD4831; Heart failure with preserved ejection fraction; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — AZD4831

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Formulation A + Formulation B) (Experimental): Participants will receive a single oral dose of Treatment 1: Formulation A followed by a washout period of at least 14 days from first dose of AZD4831. After the washout period, participants will receive a single oral dose of Treatment 2: AZD4831 Formulation B.
  Interventions: Drug: AZD4831
- Sequence 2 (Formulation B + Formulation A) (Experimental): Participants will receive a single oral dose of Treatment 2: Formulation B followed by a washout period of at least 14 days from first dose of AZD4831. After the washout period, participants will receive a single oral dose of Treatment 1 Formulation A.
  Interventions: Drug: AZD4831

INTERVENTIONS:
Drug: AZD4831 — Participants will receive a single oral dose of AZD4831 Formulation A Or a single oral dose of AZD4831 Formulation B on Day 1 Period 1. Depending on what Formulation was received on Day 1 Period 1, participants will receive either a single oral dose of AZD4831 Formulation A Or a single oral dose of AZD4831 Formulation B on Day 1 of Period 2. Each period lasts for 8 days.

SUMMARY:
A study to assess the relative bioavailability and safety of different formulations of AZD4831 in fasted state in healthy volunteers.

DETAILED DESCRIPTION:
This study will be a randomized, open-label, 2-period, 2-treatment, single-dose, single-center, crossover study conducted at a single Clinical Unit. A total of 30 healthy male and female participants will be randomized to ensure that at least 26 participants are evaluable .

The study will comprise of:

* A Screening Period of maximum 28 days.
* Period 1: single oral dose AZD4831 Formulation A or B on Day 1.
* Period 2: single oral dose AZD4831 Formulation A or B on Day 1.
* A final Follow-up Visit after the last administration of Investigational medicinal product (IMP) (14 days [+ 3 days] post final dose).

There will be a minimum washout period of at least 14 days from the first dose of AZD4831.

Participants will receive single doses of AZD4831 (2 different formulations) on 2 occasions under fasted conditions.

Participants will be given the following treatments and randomly assigned to the treatment sequence(s): AB, BA

* Treatment 1 (Reference), AZD4831 Formulation A, oral dosage form), fasted.
* Treatment 2 (Test), AZD4831 Formulation B, oral dosage from), fasted.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Male participants must adhere to the contraception methods.
* Females must have a negative pregnancy test at screening and on admission to the Clinical Unit, must not be lactating and must be of non-childbearing potential, confirmed at screening by fulfilling one of the following criteria:

  1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and Follicle-stimulating hormone (FSH) levels in the postmenopausal range.
  2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Have a Body mass index (BMI) between 18.5 and 30 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg inclusive at Screening.

Exclusion Criteria:

* Any clinically significant abnormalities on 12-lead Electrocardiogram (ECG) at the Screening Visit, as judged by the Investigator.
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP.
* History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
* Known or suspected Gilbert's syndrome.
* History or ongoing allergy/hypersensitivity to drugs (including, but not limited to rash, angioedema, acute urticaria).
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks before the first administration of AZD4831.
* Participants who previously received AZD4831.
* Any of the following signs or confirmation of COVID-19 infection:

  1. Participant has a positive SARS-CoV-2 reverse transcription-PCR test result within 2 weeks before the Screening Visit or between the Screening Visit and Randomization.
  2. Clinical signs and symptoms consistent with COVID-19 (eg, fever, dry cough, dyspnea, sore throat, fatigue) 2 weeks before the Screening Visit or between the Screening Visit and Randomization.
  3. Participant has been hospitalized with COVID-19 infection within the last 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability (Frel) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Maximum observed plasma (peak) drug concentration (Cmax) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Area under the plasma concentration-curve from zero to the last quantifiable concentration (AUClast) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Area under plasma concentration-time curve from zero to infinity (AUCinf) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Terminal rate constant, estimated by log-linear least squares regression of the terminal part of the concentration-time curve (λz) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t1/2λz) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Time of last observed (quantifiable) concentration (tlast) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Last observed (quantifiable) concentration (Clast) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | Day 1, Day 2 to Day 8 and Day 14
  The relative bioavailability of a new AZD4831 formulation compared to the formulation used in an ongoing Phase 2b study and in a couple Phase 1 studies in healthy volunteers will be evaluated.

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | From Screening until Follow up visit (At 14 days post final dose)
  The safety and tolerability of single doses of AZD4831 in healthy volunteers will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Brooklyn, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home